CLINICAL TRIAL: NCT06410586
Title: Safety and Efficacy of Integrative Korean Medicine Treatment for Children After Traffic Accident : Retrospective Chart Review Study and Survey Research
Brief Title: Integrative Korean Medicine Treatment for Pediatrics After Traffic Accident: Retrospective Chart Review Study and Survey
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2023-11
Record Dates: First submitted 2024-04-02; First posted 2024-05-13 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-05

CONDITIONS: Pediatric ALL; Traffic Accident
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective chart review study and survey research to verify the efficacy and safety of integrative Korean medicine treatment for pediatric traffic accident patients.

DETAILED DESCRIPTION:
This study is a long-term follow-up observational study targeting patients aged 0 to 6 years who visited any of the seven branches of Jaseng Hospital of Korean Medicine for outpatient and inpatient treatments after traffic accident injuries. After obtaining consent from the guardians, retrospective collection of medical records and computer data for traffic accident patients aged 0-6 will be conducted, followed by prospective surveys through Google Forms or phone interviews with the guardians. This data will be used for causal and factor analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 0 to 6 years who have visited the institution for symptoms caused by a traffic accident and have received at least one session of integrative Korean medicine treatment as inpatient or outpatient care.
2. Among the patients described in 1, those whose guardians understand the purpose and content of the research and consent to participate in the study.
3. Among the patients described in 1, those whose guardians have the communicative ability, as well as the mental and physical capacity to respond appropriately to surveys.

Exclusion Criteria:

1. Cases where only consultation was provided or only Western medical treatment was administered at our institution.
2. Other cases deemed unsuitable for study participation by the researcher.
3. Patients with a history related to the chief complaint.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 0 to 6 years who visited one of the seven branches of Jaseng Hospital of Korean Medicine for outpatient and inpatient treatments following traffic accident injuries, from January 1, 2019, to June 30, 2023, and who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | Finish survey by October 2024
  NRS uses an 11-point scale to evaluate current neck pain and radiating pain where no pain is indicated by '0', and the worst pain imaginable by '10'. NRS was assessed long term follow up.

SECONDARY OUTCOMES:
Oswestry Disability Index(ODI) | Finish survey by October 2024
  ODI is a 10-item questionnaire developed to evaluate the degree of disability for lower back pain. Each item is divided into 6 levels, and 0 to 5 points are awarded. The higher the score, the greater the degree of disability. We will conduct an validated Korean NDI questionnaire ODI was assessed long term follow up.
NDI | Finish survey by October 2024
  Functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range: 0 (better outcome) to 50 (worse outcome) In this study, the validated Korean version questionnaire will be used. NDI was assessed long term follow up.
The five level version of EuroQol-5 Dimension (EQ-5D) | Finish survey by October 2024
  EQ-5D is most widely used as a method of indirectly calculating the quality of life from various aspects. The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about) In this study, the validated Korean version questionnaire will be used. EQ-5D was assessed long term follow up.
PedsQL™ Generic Core Scales | Finish survey by October 2024
  PedsQL™ Generic Core Scales is a 21(2-4 years old), 23(5-6 years old)-item questionnaire developed to evaluate the degree of quality of life. Each item is divided into 5 levels, and 0 to 4 points are awarded. The lesser the score, the greater the quality of life. Questionnaire was assessed long term follow up.
PedsQL™ Infant Scales | Finish survey by October 2024
  PedsQL™ Generic Core Scales is a 36(0-12 months old), 45(13-24 months old)-item questionnaire developed to evaluate the degree of quality of life. Each item is divided into 5 levels, and 0 to 4 points are awarded. The lesser the score, the greater the quality of life. Questionnaire was assessed long term follow up.
Satisfaction with integrative Korean medicine survey | Finish survey by October 2024
  For patient satisfaction questionnaire, a self-developed questionnaire will be used, including which treatment was satisfied or unsatisfaide, and why. Questionnaire was assessed long term follow up.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Dr, Study Chair — Bucheon Jaseng Hospital of Korean Medicine
Locations (1):
- Bundang Jaseng Hospital of Korean Medicine, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No